CLINICAL TRIAL: NCT03830255
Title: Calcineurin Inhibitors Among Egyptian Renal Transplant Patients: a Pharmacognetic Based Study.
Brief Title: Effect of Genetic Polymorphism on Calcineurin Inhibitors Levels in Egyptian Renal Transplant Patients
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Ahmed Mohamed Ali Ismail, Lecturer Assistant at Clinical Pharmacy and Pharmacy Practice department, Misr International University
Other Study IDs: FWA000017585
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Renal Transplantation
Keywords: Renal Transplantation; Genetic Polymorphism; CYP3A5; CYP3A4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected and stored in - 80°C environment for DNA extraction by DNA extraction kit according to manufacturer recommendation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Renal Transplant patients treated with cyclosporine: Detecting the genetic polymorphism affecting cyclosporine level
- Renal Transplant patients treated with tacrolimus: Detecting the genetic polymorphism affecting tacrolimus level

SUMMARY:
Renal transplantation is the treatment of choice for patients with end-stage renal disease (ESRD). Calcineurin Inhibitors tacrolimus and cyclosporine are the principle immunosuppressive agents administered to solid organ transplant recipients to prevent and treat allograft rejection.

The aim of the present study is to detect the incidence of some selected genetic polymorphism in Egyptian renal transplant population and investigate the influence of these genetic polymorphism (SNPs )on Cyclosporine and Tacrolimus blood concentration. In addition to detect the association between these genetic polymorphism variants and patients' clinical outcome after transplantation.

DETAILED DESCRIPTION:
Tacrolimus and cyclosporine are the principle immunosuppressive agents administered to solid organ transplant recipients to prevent and treat allograft rejection.They both exert their immunosppressive action by inhibiting the calcinurein in T-lymphoctes. Subsequently,Cyclosporin and tacrolimus are both metabolic substrates for cytochrome P450 (CYP) 3A enzymes - in particular, CYP3A4 and CYP3A5 - and are transported out of cells by the P-glycoprotein (ABCB1) efflux pump. Different expression of CYP3A4, CYP3A5 and P-glycoprotein causes patient to-patient variability in the absorption, metabolism and tissue distribution of calcineurin inhibitors. This different expression is likely to be at least partially the result of mutations in the genes encoding for these enzymes and drug transporter. This may lead to variable drug concentrations within the systemic circulation and at target sites, influencing drug efficacy. Moreover, it will influence the individual's susceptibility to drug interactions and drug toxicity

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant patients.
2. Treatment with calcineurin inhibitors (CNI) either Cyclosporine (Neoral®) or Tacrolimus (Prograf®).
3. Absence of medication known to interact with CNI
4. Age18 years and more

Exclusion Criteria:

1. Patient who experience acute rejection, graft failure.
2. Medications that interact with Calcineurin Inhibitors.
3. Pregnant or nursing women.
4. Patients who decline to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal Transplant Patients
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
CYP enzymes genetic polymorphism and calcineurin inhibitors drug levels | 3 months
  Association of CP3A4 and CYP3A5 genetic polymorphism SNPs on Cyclosporine and Tacrolimus blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Magdy El Sharkawy, MD, Principal Investigator — Ain Shams University; Abdel hameed Ibrahim Mohamed Ebid, PhD, Study Director — Helwan University; Neama Lotfy, MD, Study Director — Ain sham university; Mohamed Adel, PhD, Study Director — Helwan University
Locations (1):
- Ain shams university specialized hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided